CLINICAL TRIAL: NCT04948996
Title: Effectiveness of Group Versus Individual Self-management of Depression Using a Mobile App to Increase Treatment Adherence Among Users of a University-based Helpline in the Dominican Republic.
Brief Title: Treatment of Depression Using a Mobile Application in the Dominican Republic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID, recruitment in primary care was not possible, alternative proposed hotline recruitment methods yielded population that did not meet inclusion criteria and were too acutely ill to be eligible for study.
Sponsor: Northern Illinois University (Other)
Collaborators: University Autonoma de Santo Domingo (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21MH119851-01 (NIH)
Record Dates: First submitted 2020-03-05; First posted 2021-07-02 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Depression Mild; Depression Moderate
Keywords: depression; primary care; mobile health; motivational interviewing; global health; capacity building
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- El Buen Consejo Móvil- Group (EBCM-G) (Experimental): Participants in the group condition will be placed in groups of five participants within the app. Their version of EBCM will have the functionality to connect individuals to one another via a facilitator-guided chat room (EBCM-G), where they can respond to suggested strategies within the app and communicate with each other or their facilitator guide using voice or text.
  Interventions: Behavioral: El Buen Consejo Móvil- Group (EBCM-G)
- El Buen Consejo Móvil- Individual (EBCM-I) (Active Comparator): Participants randomized to EBCM-I will receive the same program contents without the group functionality.
  Interventions: Behavioral: El Buen Consejo Móvil- Individual (EBCM-I)

INTERVENTIONS:
Behavioral: El Buen Consejo Móvil- Group (EBCM-G) — 1. Psycho-education and Information using a CBT "toolbox" approach.
  2. Self-Assessment to track, label and describe moods by daily prompts to state or text level of mood on the mood tracker ("termómetro de animo").
  3. Symptom Identification and Management: after identifying a label for type of thinking from a pull-down list, a corresponding short 1-3-minute recorded strategy such as Thought Stopping, Increasing Pleasurable Activity, Mindfulness or Priming will be provided.
  4. Monitoring of treatment engagement and response to treatment: Reminders to engage will include text messages and phone calls from the facilitator to encourage use of the app according to a scripted protocol.
  Additionally, participants in the Group Intervention will be able to communicate with and respond to one another through the group chat rooms within the app.
  Arms: El Buen Consejo Móvil- Group (EBCM-G)
Behavioral: El Buen Consejo Móvil- Individual (EBCM-I) — 1. Psycho-education and Information using a CBT "toolbox" approach.
  2. Self-Assessment to track, label and describe moods by daily prompts to state or text level of mood on the mood tracker ("termómetro de animo").
  3. Symptom Identification and Management: after identifying a label for type of thinking from a pull-down list, a corresponding short 1-3-minute recorded strategy such as Thought Stopping, Increasing Pleasurable Activity, Mindfulness or Priming will be provided.
  4. Monitoring of treatment engagement and response to treatment: Reminders to engage will include text messages and phone calls from the facilitator to encourage use of the app according to a scripted protocol.
  Arms: El Buen Consejo Móvil- Individual (EBCM-I)

SUMMARY:
The overall objective of this study is to develop a feasible and acceptable mental health app which delivers Cognitive Behavioral Therapy (CBT) for depressed patients in the Dominican Republic. This proposal meets the research objectives of NIMH in delivering mental health care to populations with low literacy, and supporting health care systems in monitoring and improving the quality of mental health. In the proposed study, the investigators will upgrade, implement, and evaluate a depression treatment app and assess trained facilitators' capacity in managing participants' depression symptoms using the app. The investigators will conduct a randomized controlled trial (RCT) among 120 participants who screen positive for mild to moderate depression or anxiety on the Patient Health Questionnaire (PHQ-9) or GAD- 7 via a university-based Covid mental health hotline. The app, El Buen Consejo Móvil (EBCM), will be downloaded to the participants' own Android phone. Participants will be randomized to receive the EBCM app with the functionality to connect individuals to one another via a facilitator-guided chat room (ECBM-G; n= 60) or to receive the same contents as an individualized facilitator-guided CBT program without the group functionality (ECBM-I; n=60).

Recruitment and mixed-methods data collection will be conducted by phone, given current circumstances surrounding the Covid-19 pandemic. Process outcomes will be evaluated for the trained facilitators. The primary outcomes for app users will be acceptability of the app and perceptions of social interactivity for those randomized to the group condition. Validated questionnaires will be administered to measure perceived emotional support, loneliness, and interactivity. Level of adherence and effectiveness, the secondary outcomes, will be assessed by frequency of interaction with the app, completion of treatment for either treatment modality, and change in depressive symptoms.

The investigators hypothesize that the use of the app for guided self-help can be enhanced through group interaction. EBCM can result in increased access to care in low-income community settings where patients are not currently receiving treatment due to logistical barriers and the stigma of seeking care in a mental health care setting.

DETAILED DESCRIPTION:
Study design:

The investigators will implement an Optimization, Effectiveness and Implementation (OEI) Hybrid Trial, based upon preliminary work. During the first six months, the investigators will upgrade and modify the mental health app, EBCM, to improve the interface and user friendliness.

Aim 1 (Optimization): Investigators will integrate app enrollment within a mental health hotline staffed by research assistants who are licensed psychologists. Protocols will be developed and produced for all hotline volunteers, including depression screening, evaluation and criteria for referral, and recruitment of individuals for study participation. Facilitators will receive extensive training for encouraging and guiding participants in usage of the app, and for facilitating chat rooms among the EBCM-G study arm. Process outcomes assessed among the app facilitators will include 1) feasibility, 2) fidelity, 3) acceptability of the training, and 4) perceived confidence in identifying and managing patients' symptoms of depression.

Aim 2 (Effectiveness and Implementation): Investigators will conduct an RCT with 120 participants who will be randomized to receive either the group treatment modality (El Buen Consejo Móvil-Group; EBCM-G) or the individual treatment modality (El Buen Consejo Móvil-Individual; EBCM-I). Participants will be followed for the duration of the 6-week intervention. Participants randomized to EBCM-G will be placed in groups of five participants within the app. Their version of the app will have the functionality to connect individuals to one another via a facilitator-guided chat room where they may respond to suggested strategies within the app and communicate with each other or their facilitator using voice or text. Participants randomized to EBCM-I will receive the same program contents without the group functionality.

Procedures:

For study recruitment, research assistants staffing the hotline will screen patients initially with the PHQ-2,and GAD-2 followed by the PHQ-9 and/or GAD-7 if positive, and will refer individuals with mild to moderate depression to the research team for an explanation of the study and the informed consent process.

Study participants will undergo baseline data collection after providing informed consent, and will then be provided with one week of prepaid internet access to allow them to download and begin using the EBCM app. Upon installing the app, participants will watch an an introductory video on how to navigate the app. After initial log-in, participants will be randomized to EBCM-G or EBCM-I using a computer-generated randomization series. After demonstrating engagement with the app during the first week, participants will receive additional prepaid internet access to continue using the app during the subsequent five weeks. EBCM will be delivered in twice daily 1-3-minute presentations.

The facilitators will undergo extensive training and will also formally consent to study participation. They will participate in mock-trials of dissemination, and interviews concerning implementation of the app. For their training in facilitation of treatment engagement, they will first receive two days of training in the scripted protocol for app coaching including the previously developed EMPDA Motivational Interviewing intervention, such as the use of supportive dialogue such as praise, reminders, non-judgmental suggestions. Facilitators will also be trained in criteria for referral in the event of symptom exacerbation or suicidal ideation as well as confidentiality and privacy during this first phase of training.

Second, the facilitators will participate in a one-week trial period of the EBCM app where supportive dialogue will be modeled by the PI's responses to comments within the app. Third, through the administration of the Internet-delivered CBT - Therapist Rating Scale (ICBT-TRS), the investigators will provide feedback to the facilitators related to their fidelity to CBT principles. During the first week, monitoring and responses will be provided on a daily basis according to a scripted protocol, while during the second and third weeks, the facilitators will review the responses to each session three times/week and offer feedback to each participant. Finally, during Weeks 4-6, participants will receive responses on a twice weekly basis. The facilitators will participate in weekly in group discussions with the PI (Dr. Susan Caplan) and Co-Investigator (Lic. Angelina Sosa Lovera) using a secure group platform to share information and reinforce best practices.

ELIGIBILITY:
Participants in Aim 1, research assistants/facilitators:

Inclusion criteria:

* Equal to or greater than age 18 years of age
* Baccalaureate degree in psychology
* Licensed as a clinical psychologist
* Able to speak and understand Spanish and read at a third grade level (for texting within the app).

Exclusion criteria:

* Age under 18 years

Participants in Aim 2, app users:

Inclusion criteria:

* Equal to or greater than age 18 years of age
* Have a positive score on the Patient Health Questionnaire (PHQ-9) of >/=5 and <15 (indicating mild to moderate depressive disorder)
* Have access to a working mobile smart phone
* Able to speak and understand Spanish and read at a third grade level (for texting within the app).

Exclusion criteria:

* age under 18 years
* PHQ-9 score < 5 or >/=15
* A history of psychiatric hospitalization for bipolar disorder, severe mental disorder, significant cognitive impairment, hearing or speech impairment, non-Spanish speaking

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Adapted Computer-Mediated Communication Questionnaire (CMCQ) | Midline (three weeks)
  Participants' perceptions of acceptability and social interactivity of the app will first be assessed at midline (three weeks after initiation of the 6-week intervention) through close-ended rating scale questions derived from the Computer-Mediated Communication Questionnaire (CMCQ). The CMCQ measures attitudes towards tech-mediated communication, consisting of four domains: social context, privacy, interactivity, and online communication (alpha coefficient of reliability = 0.83). In the present study, the adapted questions will explore these domains as they relate to app contents, engagement, mood states while using the app, and barriers and facilitators to app use. Follow-up open-ended questions will be administered alongside the close-ended questions to all participants in order to collect qualitative data that will provide context for interpreting the quantitative data.
Adapted Computer-Mediated Communication Questionnaire (CMCQ) | An average of six weeks
  Participants' perceptions of acceptability and social interactivity of the app will be assessed a second time at endline (immediately after the end of the 6-week intervention) through close-ended rating scale questions derived from the Computer-Mediated Communication Questionnaire (CMCQ). The CMCQ measures attitudes towards tech-mediated communication, consisting of four domains: social context, privacy, interactivity, and online communication (alpha coefficient of reliability = 0.83). In the present study, the adapted questions will explore these domains as they relate to app contents, engagement, mood states while using the app, and barriers and facilitators to app use. Follow-up open-ended questions will be administered to a sub-set of at least 15 participants at endline; it is anticipated that this qualitative data will provide context for interpreting the quantitative data.
Adapted Depression Training Program Evaluation (DTPE) | Through study completion; 18 months
  The facilitators' impressions of the training and the app itself will be assessed through the administration of an adapted version of the Depression Training Program Evaluation (DTPE) at the end of the intervention period. Based on the Hartford Foundation's nurse depression training program, this tool assesses feasibility of implementation, perceived acceptability of the training, perceived changes in knowledge level and confidence in one's ability to identify and manage participants' depressive symptoms, perceived changes in confidence in one's ability to communicate with participants, and perceived outcomes of the intervention for participants. In the present study, the adapted data collection instrument includes both close-ended Likert-scale rating questions as well as open-ended questions with probes.
Change in NIH Toolbox Emotional Support Scale score | At Baseline (0 weeks) and at six weeks
  Participants' perceived emotional support will be assessed at baseline (pre-intervention) and endline (post-intervention). Emotional support will be measured using the 8-item emotional support sub-scale from the validated Spanish version of the NIH Toolbox Social Relationship Scales. This sub-scale includes items related to having someone available with whom to discuss problems and who may provide empathy, support, and suggestions. The alpha coefficient of reliability for the emotional support sub-scale is 0.969. Participants rate the eight items on a five-point frequency scale (1-Never; 2-Rarely; 3-Sometimes; 4-Usually; 5-Always) over a past-month time frame. Scores may range from 8 to 40, with higher scores indicating greater levels of emotional support.
Change in Three-Item Loneliness Scale score | At Baseline (0 weeks) and at 6 weeks
  Participants' perceived loneliness will be assessed at baseline (pre-intervention) and endline (post-intervention). Perceived loneliness will be measured through the Three-item Loneliness Scale, which was derived from the R-UCLA Loneliness Scale with the goal of providing a measure that is easy to administer through telephone surveys. The Three-item Loneliness Scale has high internal consistency and an alpha coefficient of reliability of 0.72. Participants respond to three questions about perceived loneliness using a three-point frequency scale (1-Hardly ever; 2-Some of the time; and 3-Often). Scores may range from 3 to 9, with higher scores indicating greater perceived loneliness.
Adherence | Week 1
  Participant adherence to EBCM by ascertainment of number of sessions with participation (either voice or text response) divided by maximum number of sessions (10)
Adherence | Week 2
  Participant adherence to EBCM by ascertainment of number of sessions with participation (either voice or text response) divided by maximum number of sessions (20)
Adherence | Week 3
  Participant adherence to EBCM by ascertainment of number of sessions with participation (either voice or text response) divided by maximum number of sessions (30)
Adherence | Week 4
  Participant adherence to EBCM by ascertainment of number of sessions with participation (either voice or text response) divided by maximum number of sessions (40)
Adherence | Week 5
  Participant adherence to EBCM by ascertainment of number of sessions with participation (either voice or text response) divided by maximum number of sessions (50)
Adherence | Week 6
  Participant adherence to EBCM by ascertainment of number of sessions with participation (either voice or text response) divided by maximum number of sessions (60)

SECONDARY OUTCOMES:
Measure of Staff/Patient interaction scale | At six weeks
  To assess the facilitators' fidelity to and use of motivational interviewing (MI) practices, participants will complete the Measure of Staff/Patient interaction scale at endline. This 10-item scale measures the extent to which participants perceive that the facilitator is communicating in a manner that is supportive and reflective of MI principles. The scale factors align with the the three components of MI: collaboration with the client; elicitation of client's own ideas about change; and autonomy/support to encourage the patient's decision-making. The factors have alpha coefficients of reliability ranging from 0.73-0.94; the overall scale has an alpha coefficient of 0.90. The rater (i.e. the participant) rates each items on a five-point frequency scale ranging from 1-Never to 5-Always or almost always. After reverse-scoring three items, final scores may range from 10 to 50, with higher scores indicating greater levels of fidelity to MI strategies.
Internet-delivered Cognitive Behavior Therapy - Therapist Rating Scale (ICBT-TRS) | Intervention Weeks 1-6
  The Internet-delivered Cognitive Behavioral Therapy-Therapist Rating Scale (ICBT-TRS) will be employed to assess facilitator fidelity to the communication strategies delivered through the training for coaching participants. This validated behavioral checklist rates the adherence and quality of usage of specific behavior change communication strategies related to nine domains such as "Builds Rapport" and "Praises Effort." The scale has demonstrated excellent inter-rater reliability in total scores (ICC = 0.91; CI = 0.78, 0.97). For each domain, the study subject is given a rating of 0 (absence of behavior), 1 (inadequate performance/significant recommendations made), or 3 (adequate performance/minor recommendations). Scores may range from 0 to 27, with higher scores indicating increased fidelity. In the present study, the PI and co-I will use the ICBT-TRS to examine the facilitators' communication with participants throughout the intervention period.
Change in Patient Health Questionnaire (PHQ-9) score | Baseline - 0 weeks and at Week 1
  Level of depression will be assessed by the Patient Heath Questionnaire (PHQ-9), which consists of the nine criteria on which DSM-IV diagnosis of depressive disorders is based. Each of the nine items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks. A score of 5-9 indicates mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-27, severe depression. In large scale primary care studies, sensitivity was 88% and specificity was 88% for major depression at a score of greater than or equal to 10. The Spanish version has demonstrated good to excellent reliability in various Latin American countries. In the present study, the PHQ-9 will be administered on four occasions within the app (weeks 1, 2, 4, and 5) and on two occasions by phone (weeks 3 and 6). It is anticipated that a decrease of 5 points on the PHQ-9 will result from participating in the full 6-week intervention.
Change in Patient Health Questionnaire (PHQ-9) score | Baseline - 0 weeks and at Week 2
  Level of depression will be assessed by the Patient Heath Questionnaire (PHQ-9), which consists of the nine criteria on which DSM-IV diagnosis of depressive disorders is based. Each of the nine items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks. A score of 5-9 indicates mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-27, severe depression. In large scale primary care studies, sensitivity was 88% and specificity was 88% for major depression at a score of greater than or equal to 10. The Spanish version has demonstrated good to excellent reliability in various Latin American countries. In the present study, the PHQ-9 will be administered on four occasions within the app (weeks 1, 2, 4, and 5) and on two occasions by phone (weeks 3 and 6). It is anticipated that a decrease of 5 points on the PHQ-9 will result from participating in the full 6-week intervention.
Change in Patient Health Questionnaire (PHQ-9) score | Baseline - 0 weeks and at Week 3
  Level of depression will be assessed by the Patient Heath Questionnaire (PHQ-9), which consists of the nine criteria on which DSM-IV diagnosis of depressive disorders is based. Each of the nine items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks. A score of 5-9 indicates mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-27, severe depression. In large scale primary care studies, sensitivity was 88% and specificity was 88% for major depression at a score of greater than or equal to 10. The Spanish version has demonstrated good to excellent reliability in various Latin American countries. In the present study, the PHQ-9 will be administered on four occasions within the app (weeks 1, 2, 4, and 5) and on two occasions by phone (weeks 3 and 6). It is anticipated that a decrease of 5 points on the PHQ-9 will result from participating in the full 6-week intervention.
Change in Patient Health Questionnaire (PHQ-9) score | Baseline - 0 weeks and at Week 4
  Level of depression will be assessed by the Patient Heath Questionnaire (PHQ-9), which consists of the nine criteria on which DSM-IV diagnosis of depressive disorders is based. Each of the nine items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks. A score of 5-9 indicates mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-27, severe depression. In large scale primary care studies, sensitivity was 88% and specificity was 88% for major depression at a score of greater than or equal to 10. The Spanish version has demonstrated good to excellent reliability in various Latin American countries. In the present study, the PHQ-9 will be administered on four occasions within the app (weeks 1, 2, 4, and 5) and on two occasions by phone (weeks 3 and 6). It is anticipated that a decrease of 5 points on the PHQ-9 will result from participating in the full 6-week intervention.
Change in Patient Health Questionnaire (PHQ-9) score | Baseline - 0 weeks and at Week 5
  Level of depression will be assessed by the Patient Heath Questionnaire (PHQ-9), which consists of the nine criteria on which DSM-IV diagnosis of depressive disorders is based. Each of the nine items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks. A score of 5-9 indicates mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-27, severe depression. In large scale primary care studies, sensitivity was 88% and specificity was 88% for major depression at a score of greater than or equal to 10. The Spanish version has demonstrated good to excellent reliability in various Latin American countries. In the present study, the PHQ-9 will be administered on four occasions within the app (weeks 1, 2, 4, and 5) and on two occasions by phone (weeks 3 and 6). It is anticipated that a decrease of 5 points on the PHQ-9 will result from participating in the full 6-week intervention.
Change in Patient Health Questionnaire (PHQ-9) score | Baseline - 0 weeks and at Week 6
  Level of depression will be assessed by the Patient Heath Questionnaire (PHQ-9), which consists of the nine criteria on which DSM-IV diagnosis of depressive disorders is based. Each of the nine items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks. A score of 5-9 indicates mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-27, severe depression. In large scale primary care studies, sensitivity was 88% and specificity was 88% for major depression at a score of greater than or equal to 10. The Spanish version has demonstrated good to excellent reliability in various Latin American countries. In the present study, the PHQ-9 will be administered on four occasions within the app (weeks 1, 2, 4, and 5) and on two occasions by phone (weeks 3 and 6). It is anticipated that a decrease of 5 points on the PHQ-9 will result from participating in the full 6-week intervention.

OTHER OUTCOMES:
Service delivery | Baseline - Week 0
  Pre-intervention proportions of patients with MDD who are ineligible for study participation who are referred to treatment.
Change in Generalized Anxiety Disorder Scale (GAD-7) score | Baseline - 0 weeks; Week 3
  Level of anxiety will be assessed by the Generalized Anxiety Disorder Score (GAD-7) score which consists of the seven criteria on which DSM-IV diagnosis of anxiety disorders is based. Each of the seven items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks.
Change in Generalized Anxiety Disorder Scale (GAD-7) score | Baseline - 0 weeks; Week 6
  Level of anxiety will be assessed by the Generalized Anxiety Disorder Score (GAD-7) score which consists of the seven criteria on which DSM-IV diagnosis of anxiety disorders is based. Each of the seven items is scored on a three-point frequency scale ranging from 0-"not at all" to 3-"nearly every day" for the previous two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Caplan, PhD, Principal Investigator — Northern Illinois University
Locations (2):
- University of Northern Illinois, DeKalb, Illinois, United States
- University Autonoma de Santo Domingo, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
Research resources generated with funds from this grant will be freely distributed, as available, to qualified academic investigators for noncommercial research. The investigators at University of Northern Illinois and the University Autonoma de Santo Domingo, will ensure that clinical trial(s) under the award are registered and results information is submitted to ClinicalTrials.gov
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Six months after initial recruitment until 10 years after study completion
Access Criteria: Data will be shared to qualified researchers through presentations at scientific meetings, through ClinicalTrials.gov and the NIMH Database Archives following NIH guidelines. Data will be distributed without cost to approved outside collaborators under appropriate agreements for noncommercial research. Approved outside collaborators will be sponsored by an institution with an FWA assurance number, have a research-related need for the information, and certify the research need by submitting a Data Use Certification. We will make the data and associated documentation available to users only under a specific data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. No additional funds are needed for this plan.
URL: https://nda.nih.gov/get/access-data.html

REFERENCES:
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Belkin GS, Unutzer J, Kessler RC, Verdeli H, Raviola GJ, Sachs K, Oswald C, Eustache E. Scaling up for the "bottom billion": "5 x 5" implementation of community mental health care in low-income regions. Psychiatr Serv. 2011 Dec;62(12):1494-502. doi: 10.1176/appi.ps.000012011. PMID 22193798
- [Background] World Health Organization. Mental health action plan 2013-2020. Geneva, Switzerland: WHO 2013.Available at: http://apps.who.int/iris/bitstream/10665/89966/1/9789241506021_eng.pdf?ua=1
- [Background] Caplan S, Little TV, Reyna P, Sosa Lovera A, Garces-King J, Queen K, Nahar R. Mental health services in the Dominican Republic from the perspective of health care providers. Glob Public Health. 2018 Jul;13(7):874-898. doi: 10.1080/17441692.2016.1213308. Epub 2016 Aug 29. PMID 27568727
- [Background] Caplan S, Little TV, Garces-King J. Stigma about Mental Illness among Multidisciplinary Health Care Providers. International Perspectives in Psychology: Research, Practice and Consultation. 2016;5(3):196- 206 http://dx.doi.org/10.1037/ipp0000057
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Donker T, Petrie K, Proudfoot J, Clarke J, Birch MR, Christensen H. Smartphones for smarter delivery of mental health programs: a systematic review. J Med Internet Res. 2013 Nov 15;15(11):e247. doi: 10.2196/jmir.2791. PMID 24240579
- [Background] Alegria M, Mulvaney-Day N, Woo M, Torres M, Gao S, Oddo V. Correlates of past-year mental health service use among Latinos: results from the National Latino and Asian American Study. Am J Public Health. 2007 Jan;97(1):76-83. doi: 10.2105/AJPH.2006.087197. Epub 2006 Nov 30. PMID 17138911
- [Background] van Ballegooijen W, Cuijpers P, van Straten A, Karyotaki E, Andersson G, Smit JH, Riper H. Adherence to Internet-based and face-to-face cognitive behavioural therapy for depression: a meta-analysis. PLoS One. 2014 Jul 16;9(7):e100674. doi: 10.1371/journal.pone.0100674. eCollection 2014. PMID 25029507
- [Background] Andersson G, Topooco N, Havik O, Nordgreen T. Internet-supported versus face-to-face cognitive behavior therapy for depression. Expert Rev Neurother. 2016;16(1):55-60. doi: 10.1586/14737175.2015.1125783. Epub 2015 Dec 15. PMID 26610160
- [Background] Cuijpers P, Donker T, van Straten A, Li J, Andersson G. Is guided self-help as effective as face-to-face psychotherapy for depression and anxiety disorders? A systematic review and meta-analysis of comparative outcome studies. Psychol Med. 2010 Dec;40(12):1943-57. doi: 10.1017/S0033291710000772. Epub 2010 Apr 21. PMID 20406528
- [Background] Waller R, Gilbody S. Barriers to the uptake of computerized cognitive behavioural therapy: a systematic review of the quantitative and qualitative evidence. Psychol Med. 2009 May;39(5):705-12. doi: 10.1017/S0033291708004224. Epub 2008 Sep 24. PMID 18812006
- [Background] Gilbody S, Littlewood E, Hewitt C, Brierley G, Tharmanathan P, Araya R, Barkham M, Bower P, Cooper C, Gask L, Kessler D, Lester H, Lovell K, Parry G, Richards DA, Andersen P, Brabyn S, Knowles S, Shepherd C, Tallon D, White D; REEACT Team. Computerised cognitive behaviour therapy (cCBT) as treatment for depression in primary care (REEACT trial): large scale pragmatic randomised controlled trial. BMJ. 2015 Nov 11;351:h5627. doi: 10.1136/bmj.h5627. PMID 26559241
- [Background] Vis C, Mol M, Kleiboer A, Buhrmann L, Finch T, Smit J, Riper H. Improving Implementation of eMental Health for Mood Disorders in Routine Practice: Systematic Review of Barriers and Facilitating Factors. JMIR Ment Health. 2018 Mar 16;5(1):e20. doi: 10.2196/mental.9769. PMID 29549072
- [Background] Mohr DC, Burns MN, Schueller SM, Clarke G, Klinkman M. Behavioral intervention technologies: evidence review and recommendations for future research in mental health. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):332-8. doi: 10.1016/j.genhosppsych.2013.03.008. Epub 2013 May 8. PMID 23664503
- [Background] Labrique AB, Vasudevan L, Kochi E, Fabricant R, Mehl G. mHealth innovations as health system strengthening tools: 12 common applications and a visual framework. Glob Health Sci Pract. 2013 Aug 6;1(2):160-71. doi: 10.9745/GHSP-D-13-00031. eCollection 2013 Aug. PMID 25276529
- [Background] Bakker D, Kazantzis N, Rickwood D, Rickard N. Mental Health Smartphone Apps: Review and Evidence-Based Recommendations for Future Developments. JMIR Ment Health. 2016 Mar 1;3(1):e7. doi: 10.2196/mental.4984. PMID 26932350
- [Background] Caplan S, Reyna-Liberato P, Sosa Lovera A. Methodological challenges to mHealth Research in Low and Middle Income Countries: The Untold Story. Podium presentation. Eastern Nursing Research Society. Newark Liberty Marriott, Newark, NJ, April 11-13, 2018.
- [Background] Caplan S. Interprofessional Development of a Self-Guided App for Depression. National Association of Hispanic Nurses (NAHN) 42 nd Annual Conference. Phoenix, AZ, July 18- 22, 2017
- [Background] Ferrari AJ, Somerville AJ, Baxter AJ, Norman R, Patten SB, Vos T, Whiteford HA. Global variation in the prevalence and incidence of major depressive disorder: a systematic review of the epidemiological literature. Psychol Med. 2013 Mar;43(3):471-81. doi: 10.1017/S0033291712001511. Epub 2012 Jul 25. PMID 22831756
- [Background] Whiteford HA, Baxter AJ. The Global Burden of Disease 2010 Study: what does it tell us about mental disorders in Latin America? Braz J Psychiatry. 2013 Apr-Jun;35(2):111-2. doi: 10.1590/1516-4446-2012-3502. No abstract available. PMID 23904013
- [Background] Woo JM, Kim W, Hwang TY, Frick KD, Choi BH, Seo YJ, Kang EH, Kim SJ, Ham BJ, Lee JS, Park YL. Impact of depression on work productivity and its improvement after outpatient treatment with antidepressants. Value Health. 2011 Jun;14(4):475-82. doi: 10.1016/j.jval.2010.11.006. Epub 2011 Apr 22. PMID 21669372
- [Background] Cuijpers P. Prevention of depressive disorders: towards a further reduction of the disease burden of mental disorders. Early Interv Psychiatry. 2011 Aug;5(3):179-80. doi: 10.1111/j.1751-7893.2011.00282.x. No abstract available. PMID 21791028
- [Background] Bogner HR, Morales KH, Reynolds CF 3rd, Cary MS, Bruce ML. Course of depression and mortality among older primary care patients. Am J Geriatr Psychiatry. 2012 Oct;20(10):895-903. doi: 10.1097/JGP.0b013e3182331104. PMID 21997603
- [Background] Lyness JM. Naturalistic outcomes of minor and subsyndromal depression in older primary care patients. Int J Geriatr Psychiatry. 2008 Aug;23(8):773-81. doi: 10.1002/gps.1982. PMID 18200611
- [Background] Woo JM, Jeon HJ, Kim HJ, Lee KH, Lee CU, Noh JS, Lee CH, Hong JP. Excess cost of non-remission among outpatients with major depressive disorder. Int J Ment Health Syst. 2014 Nov 15;8(1):42. doi: 10.1186/1752-4458-8-42. eCollection 2014. PMID 25435902
- [Background] Weaver LJ, Mendenhall E. Applying syndemics and chronicity: interpretations from studies of poverty, depression, and diabetes. Med Anthropol. 2014;33(2):92-108. doi: 10.1080/01459740.2013.808637. PMID 24512380
- [Background] March D, Luchsinger JA, Teresi JA, Eimicke JP, Findley SE, Carrasquillo O, Palmas W. High rates of depressive symptoms in low-income urban Hispanics of Caribbean origin with poorly controlled diabetes: correlates and risk factors. J Health Care Poor Underserved. 2014 Feb;25(1):321-31. doi: 10.1353/hpu.2014.0027. PMID 24509029
- [Background] World Health Organization. (2010) mhGAP Intervention Guide. Geneva, World Health Organization, Department of Mental Health and Substance Abuse, 2010
- [Background] Piette JD, Marinec N, Gallegos-Cabriales EC, Gutierrez-Valverde JM, Rodriguez-Saldana J, Mendoz-Alevares M, Silveira MJ. Spanish-speaking patients' engagement in interactive voice response (IVR) support calls for chronic disease self-management: data from three countries. J Telemed Telecare. 2013 Feb;19(2):89-94. doi: 10.1177/1357633x13476234. Epub 2013 Mar 26. PMID 23532005
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Titov N, Andrews G, Davies M, McIntyre K, Robinson E, Solley K. Internet treatment for depression: a randomized controlled trial comparing clinician vs. technician assistance. PLoS One. 2010 Jun 8;5(6):e10939. doi: 10.1371/journal.pone.0010939. PMID 20544030
- [Background] Cuijpers P, Andersson G, Donker T, van Straten A. Psychological treatment of depression: results of a series of meta-analyses. Nord J Psychiatry. 2011 Dec;65(6):354-64. doi: 10.3109/08039488.2011.596570. Epub 2011 Jul 20. PMID 21770842
- [Background] Christensen H, Griffiths KM, Farrer L. Adherence in internet interventions for anxiety and depression. J Med Internet Res. 2009 Apr 24;11(2):e13. doi: 10.2196/jmir.1194. PMID 19403466
- [Background] Spek V, Cuijpers P, Nyklicek I, Riper H, Keyzer J, Pop V. Internet-based cognitive behaviour therapy for symptoms of depression and anxiety: a meta-analysis. Psychol Med. 2007 Mar;37(3):319-28. doi: 10.1017/S0033291706008944. Epub 2006 Nov 20. PMID 17112400
- [Background] Sander L, Rausch L, Baumeister H. Effectiveness of Internet-Based Interventions for the Prevention of Mental Disorders: A Systematic Review and Meta-Analysis. JMIR Ment Health. 2016 Aug 17;3(3):e38. doi: 10.2196/mental.6061. PMID 27535468
- [Background] Mohr DC, Lyon AR, Lattie EG, Reddy M, Schueller SM. Accelerating Digital Mental Health Research From Early Design and Creation to Successful Implementation and Sustainment. J Med Internet Res. 2017 May 10;19(5):e153. doi: 10.2196/jmir.7725. PMID 28490417
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Kelders SM, Kok RN, Ossebaard HC, Van Gemert-Pijnen JE. Persuasive system design does matter: a systematic review of adherence to web-based interventions. J Med Internet Res. 2012 Nov 14;14(6):e152. doi: 10.2196/jmir.2104. PMID 23151820
- [Background] Brouwer W, Kroeze W, Crutzen R, de Nooijer J, de Vries NK, Brug J, Oenema A. Which intervention characteristics are related to more exposure to internet-delivered healthy lifestyle promotion interventions? A systematic review. J Med Internet Res. 2011 Jan 6;13(1):e2. doi: 10.2196/jmir.1639. PMID 21212045
- [Background] Stiles-Shields C, Corden ME, Kwasny MJ, Schueller SM, Mohr DC. Predictors of outcome for telephone and face-to-face administered cognitive behavioral therapy for depression. Psychol Med. 2015 Nov;45(15):3205-15. doi: 10.1017/S0033291715001208. Epub 2015 Jun 16. PMID 26077620
- [Background] Oinas-Kukkonen H, Harjumaa M. Persuasive Systems Design: Key Issues, Process Model, and System Features. Commun Assoc Inf Syst. 2009;24(1):28.
- [Background] Alfonsson S, Olsson E, Linderman S, Winnerhed S, Hursti T. Is online treatment adherence affected by presentation and therapist support? A randomized controlled trial. Comput Hum Behav 2016 Jul;60:550- 558. [doi: 10.1016/j.chb.2016.01.035]
- [Background] Dahne J, Lejuez CW, Kustanowitz J, Felton JW, Diaz VA, Player MS, Carpenter MJ. Moodivate: A self-help behavioral activation mobile app for utilization in primary care-Development and clinical considerations. Int J Psychiatry Med. 2017 Mar;52(2):160-175. doi: 10.1177/0091217417720899. PMID 28792292
- [Background] Mohr DC, Cuijpers P, Lehman K. Supportive accountability: a model for providing human support to enhance adherence to eHealth interventions. J Med Internet Res. 2011 Mar 10;13(1):e30. doi: 10.2196/jmir.1602. PMID 21393123
- [Background] Donkin L, Christensen H, Naismith SL, Neal B, Hickie IB, Glozier N. A systematic review of the impact of adherence on the effectiveness of e-therapies. J Med Internet Res. 2011 Aug 5;13(3):e52. doi: 10.2196/jmir.1772. PMID 21821503
- [Background] Mendenhall E, De Silva MJ, Hanlon C, Petersen I, Shidhaye R, Jordans M, Luitel N, Ssebunnya J, Fekadu A, Patel V, Tomlinson M, Lund C. Acceptability and feasibility of using non-specialist health workers to deliver mental health care: stakeholder perceptions from the PRIME district sites in Ethiopia, India, Nepal, South Africa, and Uganda. Soc Sci Med. 2014 Oct;118:33-42. doi: 10.1016/j.socscimed.2014.07.057. Epub 2014 Jul 29. PMID 25089962
- [Background] Ali BS, Rahbar MH, Naeem S, Gul A, Mubeen S, Iqbal A. The effectiveness of counseling on anxiety and depression by minimally trained counselors: a randomized controlled trial. Am J Psychother. 2003;57(3):324-36. doi: 10.1176/appi.psychotherapy.2003.57.3.324. PMID 12961817
- [Background] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313
- [Background] Araya R, Rojas G, Fritsch R, Gaete J, Rojas M, Simon G, Peters TJ. Treating depression in primary care in low-income women in Santiago, Chile: a randomised controlled trial. Lancet. 2003 Mar 22;361(9362):995-1000. doi: 10.1016/S0140-6736(03)12825-5. PMID 12660056
- [Background] Winch PJ, Gilroy KE, Wolfheim C, Starbuck ES, Young MW, Walker LD, Black RE. Intervention models for the management of children with signs of pneumonia or malaria by community health workers. Health Policy Plan. 2005 Jul;20(4):199-212. doi: 10.1093/heapol/czi027. PMID 15965032
- [Background] Tripathy P, Nair N, Barnett S, Mahapatra R, Borghi J, Rath S, Rath S, Gope R, Mahto D, Sinha R, Lakshminarayana R, Patel V, Pagel C, Prost A, Costello A. Effect of a participatory intervention with women's groups on birth outcomes and maternal depression in Jharkhand and Orissa, India: a cluster-randomised controlled trial. Lancet. 2010 Apr 3;375(9721):1182-92. doi: 10.1016/S0140-6736(09)62042-0. Epub 2010 Mar 6. PMID 20207411
- [Background] Silverstein M, Diaz-Linhart Y, Cabral H, Beardslee W, Hegel M, Haile W, Sander J, Patts G, Feinberg E. Efficacy of a Maternal Depression Prevention Strategy in Head Start: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Aug 1;74(8):781-789. doi: 10.1001/jamapsychiatry.2017.1001. PMID 28614554
- [Background] Hofmann M, Broussard C, Armstrong G, Boschen MJ, Somasundaram KV. A Mental Health Training Program for Community Health Workers in India: Impact on Recognition of Mental Disorders, Stigmatizing Attitudes and Confidence. International Journal of Culture and Mental Health. 2017;10(1):62-74. http://dx.doi.org/10.1080/17542863.2016.1259340
- [Background] Moore LM, Carr A, Hartnett D. Does Group CBT for Depression Do What It Says on the Tin? A Systemic Review and Meta-analysis of Group CBT for Depressed Adults (2000-2016), Journal of Contemporary Psychotherapy. 2017; 47(3):141-157.
- [Background] Aguilera A, Garza MJ, Munoz RF. Group cognitive-behavioral therapy for depression in Spanish: culture-sensitive manualized treatment in practice. J Clin Psychol. 2010 Aug;66(8):857-67. doi: 10.1002/jclp.20706. PMID 20549680
- [Background] Marton K, Kanas N. Telehealth Modalities for Group Therapy: Comparisons to In-Person Group Therapy. Int J Group Psychother. 2016 Jan;66(1):145-150. doi: 10.1080/00207284.2015.1096109. Epub 2015 Dec 14. No abstract available. PMID 38449122
- [Background] Greene CJ, Morland LA, Macdonald A, Frueh BC, Grubbs KM, Rosen CS. How does tele-mental health affect group therapy process? Secondary analysis of a noninferiority trial. J Consult Clin Psychol. 2010 Oct;78(5):746-50. doi: 10.1037/a0020158. PMID 20873910
- [Background] Ben-Zeev D, Schueller SM, Begale M, Duffecy J, Kane JM, Mohr DC. Strategies for mHealth research: lessons from 3 mobile intervention studies. Adm Policy Ment Health. 2015 Mar;42(2):157-67. doi: 10.1007/s10488-014-0556-2. PMID 24824311
- [Background] Davidson L, Bellamy C, Guy K, Miller R. Peer support among persons with severe mental illnesses: a review of evidence and experience. World Psychiatry. 2012 Jun;11(2):123-8. doi: 10.1016/j.wpsyc.2012.05.009. PMID 22654945
- [Background] Pfeiffer PN, Heisler M, Piette JD, Rogers MA, Valenstein M. Efficacy of peer support interventions for depression: a meta-analysis. Gen Hosp Psychiatry. 2011 Jan-Feb;33(1):29-36. doi: 10.1016/j.genhosppsych.2010.10.002. Epub 2010 Nov 13. PMID 21353125
- [Background] Alegria M, Polo A, Gao S, Santana L, Rothstein D, Jimenez A, Hunter ML, Mendieta F, Oddo V, Normand SL. Evaluation of a patient activation and empowerment intervention in mental health care. Med Care. 2008 Mar;46(3):247-56. doi: 10.1097/MLR.0b013e318158af52. PMID 18388839
- [Background] Letourneau N, Secco L, Colpitts J, Aldous S, Stewart M, Dennis CL. Quasi-experimental evaluation of a telephone-based peer support intervention for maternal depression. J Adv Nurs. 2015 Jul;71(7):1587-99. doi: 10.1111/jan.12622. Epub 2015 Feb 23. PMID 25705786
- [Background] Kaplan K, Salzer MS, Solomon P, Brusilovskiy E, Cousounis P. Internet peer support for individuals with psychiatric disabilities: A randomized controlled trial. Soc Sci Med. 2011 Jan;72(1):54-62. doi: 10.1016/j.socscimed.2010.09.037. Epub 2010 Oct 26. PMID 21112682
- [Background] Takahashi Y, Uchida C, Miyaki K, Sakai M, Shimbo T, Nakayama T. Potential benefits and harms of a peer support social network service on the internet for people with depressive tendencies: qualitative content analysis and social network analysis. J Med Internet Res. 2009 Jul 23;11(3):e29. doi: 10.2196/jmir.1142. PMID 19632979
- [Background] Griffiths KM, Calear AL, Banfield M. Systematic review on Internet Support Groups (ISGs) and depression (1): Do ISGs reduce depressive symptoms? J Med Internet Res. 2009 Sep 30;11(3):e40. doi: 10.2196/jmir.1270. PMID 19793719
- [Background] Goodwin BC, Ford DE, Hsiung RC, Houston TK, Fogel J, Van Voorhees BW. First, Do No Harm: Referring Primary Care Patients with Depression to an Internet Support Group. Telemed J E Health. 2018 Jan;24(1):37-44. doi: 10.1089/tmj.2017.0004. Epub 2017 Jun 28. PMID 28657881
- [Background] Griffiths KM, Mackinnon AJ, Crisp DA, Christensen H, Bennett K, Farrer L. The effectiveness of an online support group for members of the community with depression: a randomised controlled trial. PLoS One. 2012;7(12):e53244. doi: 10.1371/journal.pone.0053244. Epub 2012 Dec 28. PMID 23285271
- [Background] Griffiths KM. Mental health Internet support groups: just a lot of talk or a valuable intervention? World Psychiatry. 2017 Oct;16(3):247-248. doi: 10.1002/wps.20444. No abstract available. PMID 28941105
- [Background] Yen C, Tu C. Multiple-group confirmatory factor analysis of the scores for online social presence: Do they measure the same thing across cultural groups? Journal of Educational Computing Research. 2011;44(2):219-242.
- [Background] Richardson JC, Swan K. Examining social presence in online courses in relation to students' perceived learning and satisfaction. Journal of Asynchronous Learning Networks. 2003;7(1):68-88.
- [Background] Russo TC, Benson S. Learning with invisible others: Online presence and its relationship to cognitive and affective learning. Educational Technology & Society. 2005;8(1):54-62.
- [Background] Caplan S. A Pilot Study of a Novel Method of Measuring Stigma about Depression Developed for Latinos in the Faith-Based Setting. Community Ment Health J. 2016 Aug;52(6):701-9. doi: 10.1007/s10597-016-0005-7. Epub 2016 Apr 16. PMID 27085546
- [Background] Caplan S, Buyske S. Depression, Help-Seeking and Self-Recognition of Depression among Dominican, Ecuadorian and Colombian Immigrant Primary Care Patients in the Northeastern United States. Int J Environ Res Public Health. 2015 Aug 27;12(9):10450-74. doi: 10.3390/ijerph120910450. PMID 26343691
- [Background] Caplan S, Cordero C. Development of a Faith-Based Mental Health Literacy Program to Improve Treatment Engagement Among Caribbean Latinos in the Northeastern United States of America. Int Q Community Health Educ. 2015;35(3):199-214. doi: 10.1177/0272684X15581347. PMID 26099153
- [Background] Caplan S, Escobar J, Paris M, Alvidrez J, Dixon JK, Desai MM, Scahill LD, Whittemore R. Cultural influences on causal beliefs about depression among Latino immigrants. J Transcult Nurs. 2013 Jan;24(1):68-77. doi: 10.1177/1043659612453745. Epub 2012 Aug 20. PMID 22913985
- [Background] Caplan S, Paris M, Whittemore R, Desai, M, Dixon J, Alvidrez J, Escobar J, Scahill LD. Correlates of Religious, Supernatural and Psychosocial Causal Beliefs about Depression among Latino Immigrants in Primary Care. Mental Health, Religion and Culture. 2010;13 (7):1469-9737, DOI: 10.1080/13674676.2010.497810
- [Background] Nuevo R, Lehtinen V, Reyna-Liberato PM, Ayuso-Mateos JL. Usefulness of the Beck Depression Inventory as a screening method for depression among the general population of Finland. Scand J Public Health. 2009 Jan;37(1):28-34. doi: 10.1177/1403494808097169. PMID 19141552
- [Background] Cayetano C, Sosa A, González R. Observatorio subregional de la conducta suicida para Centroamérica y la República Dominicana in Organización Panamericana de la Salud. Prevención de la conducta suicida. Washington, DC : OPS, 2016. [Cayetano, C. Sosa, A. & González, R Subregional suicide observatory for Central America and the Dominican Republic in Panamercan Health Organization. Prevention of suicidal behavior ISBN: 978-92-75-11919-8
- [Background] Canario Guzman JA, Espinal R, Baez J, Melgen RE, Rosario PAP, Mendoza ER. Ethical challenges for international collaborative research partnerships in the context of the Zika outbreak in the Dominican Republic: a qualitative case study. Health Res Policy Syst. 2017 Sep 25;15(1):82. doi: 10.1186/s12961-017-0246-0. PMID 28946911
- [Background] Canario JA, Lizardo J, Espinal R, Colome M. Gaps in health research in the Dominican Republic. Rev Panam Salud Publica. 2016 Apr;39(4):179-85. PMID 27657182
- [Background] Winch PJ, Leban K, Casazza L, Walker L, Pearcy K. An implementation framework for household and community integrated management of childhood illness. Health Policy Plan. 2002 Dec;17(4):345-53. doi: 10.1093/heapol/17.4.345. PMID 12424206
- [Background] Rahman SM, Ali NA, Jennings L, Seraji MH, Mannan I, Shah R, Al-Mahmud AB, Bari S, Hossain D, Das MK, Baqui AH, El Arifeen S, Winch PJ. Factors affecting recruitment and retention of community health workers in a newborn care intervention in Bangladesh. Hum Resour Health. 2010 May 3;8:12. doi: 10.1186/1478-4491-8-12. PMID 20438642
- [Background] Hoover DR. Clinical trials of behavioural interventions with heterogeneous teaching subgroup effects. Stat Med. 2002 May 30;21(10):1351-64. doi: 10.1002/sim.1139. PMID 12185889
- [Background] Podium Presentation. Tariana V. Little, Susan Caplan, Angelina Sosa Lovera, Patricia Reyna, Pak Chau, Adrian Aguilera, Jenny Ariannly Sánchez Castillo, Ester R. Shapiro. Mobile App to Prevent Depression in the Dominican Republic. Sociocultural Adaptations. Sigma Theta Tau International, Dublin, Ireland, Sunday, 30 July 2017: 11:15 AM
- [Background] Muñoz RF, Ghosh Ippen, C, Rao S, Le HL, Dwyer EV. Manual de terapia de grupo para el tratamiento cognitivo-conductual de la depresión [Healthy management of reality: group cognitive behavioral therapy manual]: Aprendiendo a manejar su realidad personal. 2000.
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Bird VJ, Le Boutillier C, Leamy M, Williams J, Bradstreet S, Slade M. Evaluating the feasibility of complex interventions in mental health services: standardised measure and reporting guidelines. Br J Psychiatry. 2014;204:316-21. doi: 10.1192/bjp.bp.113.128314. Epub 2013 Dec 5. PMID 24311549
- [Background] Hadjistavropoulos HD, Schneider LH, Klassen K, Dear BF, Titov N. Development and evaluation of a scale assessing therapist fidelity to guidelines for delivering therapist-assisted Internet-delivered cognitive behaviour therapy. Cogn Behav Ther. 2018 Nov;47(6):447-461. doi: 10.1080/16506073.2018.1457079. Epub 2018 Apr 25. PMID 29693533
- [Background] Hohman M, Matulich W. Initial validation of the motivational interviewing measure of staff interaction. Alcoholism Treatment Quarterly.2010;28(2):230-238.
- [Background] Smith M, Johnson KM, Seydel LL, Buckwalter KC. Depression training for nurses: Evaluation of an innovative program. Res Gerontol Nurs. 2010 Jul;3(3):162-75. doi: 10.3928/19404921-20100527-99. Epub 2010 Jun 30. PMID 20635801
- [Background] Agarwal S, LeFevre AE, Lee J, L'Engle K, Mehl G, Sinha C, Labrique A; WHO mHealth Technical Evidence Review Group. Guidelines for reporting of health interventions using mobile phones: mobile health (mHealth) evidence reporting and assessment (mERA) checklist. BMJ. 2016 Mar 17;352:i1174. doi: 10.1136/bmj.i1174. No abstract available. PMID 26988021
- [Background] Tu C-H. The Measurement of Social Presence in an Online Learning Environment. International Journal on E-Learning. 2002;1(2): 34-45. Norfolk, VA: Association for the Advancement of Computing in Education (AACE).
- [Background] Nick EA, Cole DA, Cho SJ, Smith DK, Carter TG, Zelkowitz RL. The Online Social Support Scale: Measure development and validation. Psychol Assess. 2018 Sep;30(9):1127-1143. doi: 10.1037/pas0000558. Epub 2018 May 21. PMID 29781664
- [Background] Procidano ME, Heller K. Measures of perceived social support from friends and from family: three validation studies. Am J Community Psychol. 1983 Feb;11(1):1-24. doi: 10.1007/BF00898416. PMID 6837532
- [Background] Khelladi Y. Case Study: Dominican Republic Alliance for Affordable Internet, February 2015. Retrieved from www.a4ai.org
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] Baca E, Saiz J, Aguera L, Caballero L, Fernandez-Liria A, Ramos J, Gil A, Madrigal M, Porras A. [Validation of the Spanish version of PRIME-MD: a procedure for diagnosing mental disorders in primary care]. Actas Esp Psiquiatr. 1999 Nov-Dec;27(6):375-83. Spanish. PMID 10611561
- [Background] Sosa, A., Tejeda, E. P[erez, W. (2018). Depression on Primary Attention, Santo Domingo Este, 2017. Presented at National Conference of Epidemiology, Santo Domingo, Dominican Republic.
- [Background] van der Feltz-Cornelis CM, Nuyen J, Stoop C, Chan J, Jacobson AM, Katon W, Snoek F, Sartorius N. Effect of interventions for major depressive disorder and significant depressive symptoms in patients with diabetes mellitus: a systematic review and meta-analysis. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):380-95. doi: 10.1016/j.genhosppsych.2010.03.011. Epub 2010 May 15. PMID 20633742
- [Background] de Jonge P, Hadj FB, Boffa D, Zdrojewski C, Dorogi Y, So A, Ruiz J, Stiefel F. Prevention of major depression in complex medically ill patients: preliminary results from a randomized, controlled trial. Psychosomatics. 2009 May-Jun;50(3):227-33. doi: 10.1176/appi.psy.50.3.227. PMID 19567761
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Braun, V. & Clark, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3, 77-101.
- [Background] Cohen, Jacob (1988). Statistical Power Analysis for the Behavioral Sciences. Routledge. ISBN 1-134- 74270-3.
- [Background] Schoenfeld D. Statistical considerations for pilot studies. Int J Radiat Oncol Biol Phys. 1980 Mar;6(3):371-4. doi: 10.1016/0360-3016(80)90153-4. No abstract available. PMID 7390914
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794
- [Background] Pan W. Sample size and power calculations with correlated binary data. Control Clin Trials. 2001 Jun;22(3):211-27. doi: 10.1016/s0197-2456(01)00131-3. PMID 11384786
- [Background] Xue X, Hoover DR. Statistical methods in cancer epidemiological studies. Methods Mol Biol. 2009;471:239-72. doi: 10.1007/978-1-59745-416-2_13. PMID 19109784
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Cesana BM, Antonelli P. Sample size calculations in clinical research should also be based on ethical principles. Trials. 2016 Mar 18;17(1):149. doi: 10.1186/s13063-016-1277-5. PMID 26993625
- [Background] Lee EC, Whitehead AL, Jacques RM, Julious SA. The statistical interpretation of pilot trials: should significance thresholds be reconsidered? BMC Med Res Methodol. 2014 Mar 20;14:41. doi: 10.1186/1471-2288-14-41. PMID 24650044
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Background] Viechtbauer W, Smits L, Kotz D, Bude L, Spigt M, Serroyen J, Crutzen R. A simple formula for the calculation of sample size in pilot studies. J Clin Epidemiol. 2015 Nov;68(11):1375-9. doi: 10.1016/j.jclinepi.2015.04.014. Epub 2015 Jun 6. PMID 26146089
- [Background] Cyranowski JM, Zill N, Bode R, Butt Z, Kelly MA, Pilkonis PA, Salsman JM, Cella D. Assessing social support, companionship, and distress: National Institute of Health (NIH) Toolbox Adult Social Relationship Scales. Health Psychol. 2013 Mar;32(3):293-301. doi: 10.1037/a0028586. PMID 23437856
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- See also: VoiceThread, LLC. (2016) — http://voicethread.com/
- See also: Digital In 2018 in the Caribbean: Essential Insights Into Internet, Social Media, Mobile, And Ecommerce Use Across The Region Part 1:West — https://www.Slideshare.Net/Wearesocial/Digital-In-2018-In-The-Caribbean-Part-1-West-86863340
- See also: The MacArthur Foundation. Depression Management Tool Kit. The John D. & Cather T. MacArthur Foundation's Initiative on Depression and Primary Care 2009 — https://www.depression-primarycare.org/clinicians/toolkits/